CLINICAL TRIAL: NCT06862973
Title: Comparison of Occlusal Force Distribution and Digital Occlusal Analysis Methods of Single Posterior Implant Restorations and Digital Occlusal Analysis Methods
Brief Title: Digital Analysis of Occlusal Force Distribution in Single-Tooth Implant Restorations
Status: Completed | Type: Observational
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, Mehmet Gözen, DDS, Department of Prosthodontics, Faculty of Dentistry, Konya Necmettin Erbakan Üniversitesi
Other Study IDs: 20754
Record Dates: First submitted 2025-03-05; First posted 2025-03-07 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-01

CONDITIONS: Occlusal Analysis
Keywords: Occlusion; Dental Implant; Occlusal Analysis; OccluSense; Medit i700
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Digital Occlusal Analysis Using Medit i700 and OccluSense in Single-Tooth Implant Restorations — This study differs from other research through the comparison of two advanced digital occlusal analysis methods-OccluSense system and MEDIT i700 intraoral scanner-to measure occlusal force distribution both before and after the insertion of single-tooth implant restorations in the posterior segment. Unlike research based upon the use of articulation paper, this study employs pressure-sensitive sensor technology (OccluSense) and scanner-based occlusion analysis (MEDIT i700) to quantitatively measure occlusal contacts and force intensity using CloudCompare and ImageJ. With the analysis of the variations that take place within the pre-and-post implant occlusion, the study provides an understanding of occlusal adaptation and how to optimize occlusal adjustments to prevent implant overload and complications, differing from the research that has previously lacked both digital force mapping and longitudinal occlusal analysis.

SUMMARY:
This study will explore the impact of single tooth implant restorations upon occlusal force distribution and the accuracy of several digital analysis methods. The biomechanical behavior of implant-supported prostheses differs from that of natural teeth, and the distribution and modulation of occlusal forces are unpredictable.

The research used the Medit i700 intraoral scanner and the OccluSense system to take pre- and post-implant measurements. The research aims to determine: How are the techniques different in the registration of occlusal contacts and force magnitude? and How does occlusal balance shift following the placement of an implant? The research findings can be used to provide clinical recommendations to optimize occlusal balancing during implant prosthetics.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 and over
* Patients with good periodontal health
* Patients with a Class I bite
* Patients with a single tooth deficiency in the posterior region planned for rehabilitation with an implant-supported single crown restoration

Exclusion Criteria:

* History of temporomandibular joint disease
* Acute pain or signs of occlusal dysfunction
* Restricted mouth opening
* Absence of a tooth distal to the planned restoration
* Occlusion instability due to prior orthodontic or surgical treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: he study population consists of adult patients requiring single posterior implant-supported restorations at Necmettin Erbakan University Faculty of Dentistry. Participants are selected based on specific inclusion criteria, including good periodontal health, a single missing tooth in the posterior region, and stable occlusion (Class I bite). Patients with a history of temporomandibular joint disorders, acute pain, occlusal dysfunction, restricted mouth opening, or prior orthodontic or surgical treatments affecting occlusion are excluded. The study aims to assess occlusal force distribution changes in a clinically relevant population undergoing implant rehabilitation, providing insights into post-restorative occlusal adjustments.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Occlusal Force Distribution from Pre-Implant to Post-Implant Restoration as Measured by Medit i700 and OccluSense | From pre-implant assessment to 2 week after final implant restoration placement.
  Occlusal force distribution was measured before and after single-tooth implant restoration using two digital occlusal analysis methods: Medit i700 intraoral scanner and OccluSense pressure sensor system. Measurements were taken under standardized conditions, ensuring maximum intercuspation position. Medit i700 provided contact area data through intraoral scans, analyzed with CloudCompare software, while OccluSense recorded occlusal force intensity and distribution, analyzed with ImageJ software. The percentage change in occlusal contact areas and force distribution was calculated between the pre- and post-implant conditions. A statistically significant change (p < 0.05) indicates an alteration in occlusal balance following the restoration.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
yes, all IPD that underlie results in a publication
Supporting Information: CSR
Time Frame: April 2025-January 2026

REFERENCES:
- [Derived] Gozen M, Guntekin N. Comparison of occlusal force distribution and digital occlusal analysis methods of single posterior implant restorations: an in vivo study. BMC Oral Health. 2025 May 26;25(1):795. doi: 10.1186/s12903-025-06205-w. PMID 40420258